CLINICAL TRIAL: NCT07261904
Title: Prospective, Observational, Multicentre, Single Group, Open-label Study to Confirm the Safety and Effectiveness of BIOCHROMADERM® Ink for the Reconstruction of the Nipple-areola Complex in Patients Undergoing Breast Reconstructive Surgery Following Mastectomy
Brief Title: BIOCHROMADERM® PMCF STUDY
Status: Recruiting | Type: Observational
Sponsor: Laboratoires BIOTIC Phocea (Industry)
Collaborators: Clinical Research Consultants, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ID-RCB 2024-A01845-42
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Reconstruction of the Nipple-areola Complex in Patients Undergoing Breast Reconstructive Surgery Following Mastectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to:

* To confirm the continued performance of BIOCHROMADERM® in restoring a near-normal pigmentary appearance of the nipple-areola complex at 3 months post-pigmentation;
* To confirm the continued safety of BIOCHROMADERM®,
* To confirm adequate usability and describe the optimal process for BIOCHROMADERM® implantation
* To assess the long-term performance of BIOCHROMADERM® in restoring a near-normal pigmentary appearance of the nipple-areola complex at 12 months post-pigmentation (Likert scale)
* To assess the evolution of performance (Likert scale) between baseline, 3 months and 12 months post-pigmentation
* To assess fading (pigment retention potential) over 12 months
* To assess the number of pigmentation adjustments needed per patient throughout the study duration
* To assess patient's satisfaction/self-confidence evolution post-treatment, both in terms of general breast appearance and as to the specific dermo-pigmentation stage
* To assess the correlation of the esthetic satisfaction/self-confidence questionnaire outcomes with those of the Likert Scale and patient satisfaction VAS at 3 months and 12 months post-pigmentation

ELIGIBILITY:
Inclusion Criteria:

* Female or male ≥18 years old,
* Requiring the reconstruction of the nipple-areola complex following mastectomy,
* Affiliated or beneficiary of a social security scheme,
* Able and willing to provide written informed consent to study participation.

Exclusion Criteria:

* Known allergy to pigment ingredients
* Active, recent or prior history of skin disease, chronic skin disease, history of hypertrophic scars, skin infection or skin inflammatory disease,
* Patients carrying a prosthesis (especially cardiac),
* Patients presenting with a coagulation disorder,
* Patients scheduled for an MRI within 6 months following pigmentation,
* Patients scheduled for a skin esthetic treatment close to the pigmentation zone (laser, peeling, abrasion, ...) shortly after pigmentation,
* Existing medical condition or organ pathology close to the skin that the Investigator considers may put the patient at risk or compromise their participation in the study,
* Pregnant or breastfeeding female,
* Currently participating to another clinical trial or having participated to a prior clinical trial within 1 month prior to inclusion into the present one,
* Personal strong objection to medical tattooing,
* Psychiatric illness/social situations that would limit ability to consent and/or to compliance with study requirements,
* Under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.

Note: The recent use of permanent wrinkle or lip filling products close to the scheduled pigmentation zone (silicon, PTFE, ...) is a contraindication in the approved product IFU but is not relevant to the breast reconstruction indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients requiring the correction of skin pigmentation in the NAC area as a result of breast reconstructive surgery following mastectomy.
  Up to 115 patients will be included into the study by 3 clinical sites, in order to obtain 103 treated patients followed up over 12 months post-procedure per protocol
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-10-12 (Estimated); Study Completion 2027-06-12 (Estimated)

PRIMARY OUTCOMES:
To confirm the continued performance of BIOCHROMADERM® in restoring a near-normal pigmentary appearance of the nipple-areola complex at 3 months post-pigmentation | 3 months post-pigmentation

SECONDARY OUTCOMES:
To confirm the continued safety of BIOCHROMADERM® | 12 months
To confirm adequate usability and describe the optimal process for BIOCHROMADERM® implantation | 12 months
To assess the long-term performance of BIOCHROMADERM® in restoring a near-normal pigmentary appearance of the nipple-areola complex at 12 months post-pigmentation (Likert scale) | 12 months
To assess the evolution of performance (Likert scale) between baseline, 3 months and 12 months post-pigmentation | 12 months
To assess fading (pigment retention potential) over 12 months | 12 months
To assess the number of pigmentation adjustments needed per patient throughout the study duration | 12 months
To assess patient's satisfaction/self-confidence evolution post-treatment, both in terms of general breast appearance and as to the specific dermo-pigmentation stage | 12 months
To assess the correlation of the esthetic satisfaction/self-confidence questionnaire outcomes with those of the Likert Scale and patient satisfaction VAS at 3 months and 12 months post-pigmentation | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Oscar Lambret, Lille
  - Hôpital de La Conception, Marseille
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No